CLINICAL TRIAL: NCT05761327
Title: Investigation of the Effects of Curcumin and Resveratrol Supplements Added to the Mediterranean Diet on Disease Severity and Inflammatory Biomarkers in Patients With Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ardahan University (Other)
Responsible Party: Principal Investigator, Özge EROL DOĞAN, Master of Science, Lecturer., Ardahan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/24
Record Dates: First submitted 2023-02-11; First posted 2023-03-09 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Mediterranean diet; Curcumin; Resveratrol; inflammatory bowel disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: Intervention Group 1: Mediterranean Diet Intervention Group 2: Mediterranean Diet + Curcumin Supplementation Intervention Group 3: Mediterranean Diet + Resveratrol Supplementation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mediterranean Diet (Active Comparator): The individuals in this group will be given a nutrition model in accordance with the Mediterranean Nutrition Program under the supervision of a dietitian for 8 weeks. Individuals will be informed about the Mediterranean diet, their questions will be answered, the current food consumption record will be examined by the dietitian and they will be asked to follow the nutrition program prepared in the most appropriate way (by considering energy, nutrient requirements and nutritional habits). Every 15 days, the nutrition program will be updated with the meetings to be made by the dietitian and the patient, and the applicability of the program will be checked through daily communication.
  Interventions: Other: Mediterranean Diet
- Curcumin Supplementation (Experimental): In addition to the Mediterranean Diet program in the 1st group for individuals in this group; 800 mg of curcumin supplement (VeNatura Curcumin Supplementary Food, Vefa, Istanbul, Turkey) will be given as 1 capsule each in the morning and evening meals.
  Interventions: Other: Mediterranean Diet; Dietary Supplement: Curcumin Supplementation
- Resveratrol Supplementation (Experimental): In addition to the Mediterranean Diet in the 1st group for individuals in this group; 250 mg resveratrol supplement (VeNatura Resveratrol Supplementary Food, Vefa, Istanbul, Turkey) will be given as 1 capsule each in the morning and evening meals.
  Interventions: Other: Mediterranean Diet; Dietary Supplement: Resveratrol Supplementation

INTERVENTIONS:
Other: Mediterranean Diet — In the Mediterranean diet; The frequency of consumption of foods such as olive oil, olives, nuts, fish, vegetables and fruits will be given in accordance with the Mediterranean diet pyramid. During the study, it is planned to develop new recipes suitable for the nutritional habits of the individual. The researcher will be able to reach the researcher 7/24 in case of any problem experienced by the individual, and the participant's questions will be answered. Nutrition counseling to this group will be supported by an oral explanation given by the dietitian.
Dietary Supplement: Curcumin Supplementation — Participants will take a daily supplement of 1600 mg of curcumin. It is planned that the participants will use 120 capsules of curcumin supplement during the research.
  Arms: Curcumin Supplementation
Dietary Supplement: Resveratrol Supplementation — Participants will take a 500mg resveratrol supplement daily. Participants are planned to use 120 capsules of resveratrol supplement during the study.
  Arms: Resveratrol Supplementation

SUMMARY:
The aim of the study was to examine and compare the effects of Mediterranean diet, curcumin supplementation with Mediterranean diet in individuals with ulcerative colitis, and resveratrol supplementation with Mediterranean diet in individuals with ulcerative colitis, on disease symptoms, quality of life, and inflammatory biomarkers.

DETAILED DESCRIPTION:
In the light of the information in the literature, it is seen that the level of evidence in the existing literature is insufficient with the data obtained in terms of dietary approaches and nutritional supplements to be applied to individuals with Ulcerative Colitis (UC). In addition, when the literature was examined, no randomized controlled study was found that specifically examined the effects of the Mediterranean diet and nutritional supplements combined with diet in individuals with UC, and also compared the effects of two different nutritional supplements applied in combination with diet. In this direction, the aims of this research are;

* Mediterranean diet in individuals with UC,
* Curcumin supplement taken together with the Mediterranean diet in individuals with UC,
* Resveratrol supplement taken with the Mediterranean diet in individuals with UC, To examine and compare their effects on disease symptoms, quality of life and inflammatory biomarkers.

Hypotheses of the Research;

H0a: Mediterranean diet has no effect on disease symptoms, quality of life an inflammatory biomarkers in individuals with UC.

H0b: Curcumin supplementation in addition to the Mediterranean diet has no effect on disease symptoms, quality of life, and inflammatory biomarkers in individuals with UC.

H0c: Resveratrol supplementation in addition to the Mediterranean diet has no effect on disease symptoms, quality of life and inflammatory biomarkers in individuals with UC.

H0d: Three approaches including Mediterranean diet, curcumin and resveratrol supplements applied in addition to diet in individuals with UC; compared to each other in terms of disease symptoms, quality of life, and inflammatory biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged >18 years,
* Those previously diagnosed with ulcerative colitis and/or newly diagnosed with clinical course, consistent histology and endoscopy by a gastroenterologist,
* Mild and Moderate activity disease was confirmed by the Truelove-Witts Severity Index,
* Using a fixed dose of 5 - aminosalicylic acid (mesalazine) and/or azathioprine,
* Who did not receive nutrition therapy in the last 3 months,
* Not using anti-inflammatory drugs and antibiotic drugs in the last 4 weeks,
* Not using curcumin and resveratrol supplements before participating in the study,
* Agreeing to participate in the study voluntarily,

Exclusion Criteria:

* Women during pregnancy or lactation
* Not meeting the inclusion criteria,
* History of chronic disease (such as diabetes), hypothyroidism and hyperthyroidism, liver, kidney and cardiovascular diseases, polycystic ovary syndrome and Cushing's syndrome,
* Taking one of the anti-inflammatory and antibiotic drugs,

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2023-02-18 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Inflammatory Bowel Disease Questionnaire (IBDQ) | Change from baseline Inflammatory Bowel Disease Questionnaire total score at 8 weeks
  The questionnaire consists of 32 questions and 4 subsections. These sections are; systemic symptoms (5 questions), emotional function (12 questions), social function (5 questions) and intestinal symptoms (10 questions). The questionnaire consists of a 7-point Likert scale system. For each question, 1 point indicates the highest level of exposure, and 7 indicates that there is no problem. Scores range from 32 to 224, with a higher score associated with higher quality of life. Turkish version of IBDQ will be used to assess patients' quality of life.
Mediterranean Diet Assessment Tool (14-MEDAS) | Change from baseline Mediterranean Diet Assessment Tool total score at 8 weeks
  The Mediterranean Diet Assessment Tool will be used to measure the adherence of the participants to the Mediterranean diet. In the 14-question scale, 1 or 0 points are taken for each question asked according to the amount of consumption and these points are added. Scores are evaluated as ≤5 (low ), 6-9 (moderate), and ≥10 (high agreement).

SECONDARY OUTCOMES:
36-Item Short Form Survey (SF-36) | Change from baseline physical function, physical role limitation, pain, general health, vitality, social function, emotional role limitation, and mental health scores at 8 weeks
  It is the most frequently used quality of life scale in the medical field and consists of 8 sub-parameters with a total of 36 items that evaluate physical and mental health. These sub-parameters are physical function, physical role limitation, pain, general health, vitality, social function, emotional role limitation, and mental health. The scores range from 0-100, with 100 points indicating the best health condition and 0 points the worst health condition.
Truelove-Witts Severity Index | Change from baseline Truelove-Witts Severity Index score at 8 weeks
  Truelove-Witts Severity Index is a clinical classification categorizes the disease as mild, moderate, and severe, based on a combination of clinical and laboratory parameters, including bowel movements, rectal bleeding, fever, tachycardia, anemia, and increased sedimentation. The Truelove-Witts classification, using clinical symptoms, is applicable to patients with ulcerative colitis,and it is easy and reliable to use in the clinic.
Body Mass Index | Change from baseline BMI at 8 weeks
  Body weight measurements and height of the volunteers will be taken with height meter and scale. All measurements will be taken in light clothing and without shoes, according to International Standards for Anthropometric Assessment (ISAK) guidelines. Body mass index (BMI) will be calculated with weight (kg) / height (m)^2 formula. Results will be interpreted as kg/m^2.
Waist Hip Circumference Ratio | Change from baseline Waist hip circumference ratio at 8 weeks
  Non-stretchable tape measure will be used for waist and hip circumference. All measurements will be taken in light clothing and without shoes, according to International Standards for Anthropometric Assessment (ISAK) guidelines. Waist hip circumference ratio will be calculated with waist circumference (cm) / hip circumference (cm).
Daily energy intake | Change from baseline from the daily energy intake at 8 weeks
  Food frequency will be evaluated by The Turkish Ministry of Health version of Food Frequency Questionnaire (FFQ). FFQ is a limited check list of foods and beverages with a frequency response section for subjects to report how often each item was consumed over the last three months. Food Record (FR) will be evaluated dietary recall. The patient will be asked to note down the foods she consumes for last 3 days. The obtained data from FFQ and FR will be entered into the BeBiS 7.1 software (BeBiS Comp., Istanbul, Turkey) and the daily energy intake(kcal) will be calculated.
Daily protein, fat, carbohydrate and fiber intake | Change from baseline from the daily protein, fat, carbohydrate and fiber intake at 8 weeks
  Food frequency will be evaluated by The Turkish Ministry of Health version of Food Frequency Questionnaire (FFQ). FFQ is a limited check list of foods and beverages with a frequency response section for subjects to report how often each item was consumed over the last three months. Food Record (FR) will be evaluated dietary recall. The patient will be asked to note down the foods she consumes for last 3 days. The obtained data from FFQ and FR will be entered into the BeBiS 7.1 software (BeBiS Comp., Istanbul, Turkey) and the daily protein, fat, carbohydrate, fiber (gram) intake will be calculated.
Daily vitamin and mineral intake (mg) | Change from baseline from the daily vitamin and mineral intake (mg) at 8 weeks
  Food frequency will be evaluated by The Turkish Ministry of Health version of Food Frequency Questionnaire (FFQ). FFQ is a limited check list of foods and beverages with a frequency response section for subjects to report how often each item was consumed over the last three months. Food Record (FR) will be evaluated dietary recall. The patient will be asked to note down the foods she consumes for last 3 days. The obtained data from FFQ and FR will be entered into the BeBiS 7.1 software (BeBiS Comp., Istanbul, Turkey) and the daily vitamin (E, B1, B2, niacin, C) and mineral (sodium, potassium, magnesium, phosphorus, iron, zinc) (mg) intake will be calculated.
Daily vitamin and mineral intake (mcg) | Change from baseline from the daily vitamin and mineral intake (mcg) at 8 weeks
  Food frequency will be evaluated by The Turkish Ministry of Health version of Food Frequency Questionnaire (FFQ). FFQ is a limited check list of foods and beverages with a frequency response section for subjects to report how often each item was consumed over the last three months. Food Record (FR) will be evaluated dietary recall. The patient will be asked to note down the foods she consumes for last 3 days. The obtained data from FFQ and FR will be entered into the BeBiS 7.1 software (BeBiS Comp., Istanbul, Turkey) and the daily vitamin (A, D, K, Folate, B12) and mineral (iodine) (mcg) intake will be calculated.
24 Hour Recall Physical Activity Record | Pre-intervention: Beginning of the study
  Individuals who will participate in the research will be asked to record the physical activities they have done within 24 hours, in minutes, and to bring them to the week in which nutritional counseling will begin. Thus, after anthropometric measurements are made on the individuals, the resting metabolic rate (RMH) will be calculated with the Harris Benedict equation and the total energy requirements will be determined together with the physical activity coefficient found by using the 24-hour physical activity record.
C-Reactive Protein | Change from baseline C-Reactive Protein (mg/dL) at 8 weeks.
  The blood tests were performed during routine controls. The C-Reactive Protein (mg/dL) biomarkers parameters to be examined.
Hemoglobin | Change from baseline hemoglobin (g/dL) at 8 weeks.
  The blood tests were performed during routine controls. The Hemoglobin (g/dL) to be examined.
Mean Corpuscular Hemoglobin | Change from baseline Mean Corpuscular Hemoglobin (pg) at 8 weeks.
  The blood tests were performed during routine controls. The Mean Corpuscular Hemoglobin (pg) parameter to be examined.
Mean Platelet Volume and Platelet Distribution Width (fL) | Change from baseline Mean Platelet Volume and Platelet Distribution Width (fL) at 8 weeks.
  The blood tests were performed during routine controls. The blood biomarkers parameters to be examined are as follows:
  Mean Platelet Volume (fL) Platelet Distribution Width (fL) All blood biomarkers will be interpret separately.
Erythrocyte Sedimentation Rate (mm/hour) | Change from baseline Erythrocyte Sedimentation Rate (mm/hour) at 8 weeks.
  The blood tests were performed during routine controls. The blood biomarkers parameters to be examined are as follows:
  Erythrocyte Sedimentation Rate (mm/hour)
White blood cell and Thrombocyte (10^3/uL) | Change from baseline White blood cell and Thrombocyte (10^3/uL) at 8 weeks.
  The blood tests were performed during routine controls. The blood biomarkers parameters to be examined are as follows:
  White blood cell (10^3/uL) Thrombocyte (10^3/uL) All blood biomarkers will be interpret separately.
Blood biomarkers (%) | Change from baseline blood parameters (%) at 8 weeks.
  The blood tests were performed during routine controls. The blood biomarkers parameters to be examined are as follows:
  Hematocrit (%) Pro-calcitonin (%) Lymphocyte (%) Monocyte (%) Neutrophil (%) Eosinophil (%) Basophil (%) Immune Globulin G (%) Platelet-Large cell ratio (%) Red Cell Distribution Width (%)

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Inonu University Turgut Ozal Medical Center, Malatya
  - Malatya Training and Research Hospital, Malatya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Judge TA LG. Inflammatory Bowel Disease. In: Friedman SL MK, Grendell JH, editor. CURRENT Diagnosis&Treatment in Gastroenterology 2th ed. America: McGraw-Hill Companies; 2003.
- [Background] Sands BE. From symptom to diagnosis: clinical distinctions among various forms of intestinal inflammation. Gastroenterology. 2004 May;126(6):1518-32. doi: 10.1053/j.gastro.2004.02.072. No abstract available. PMID 15168364
- [Background] Kothari M, Mudireddy P, Swaminath A. Patient considerations in the management of ulcerative colitis - role of vedolizumab. Ther Clin Risk Manag. 2015 Aug 19;11:1235-42. doi: 10.2147/TCRM.S65650. eCollection 2015. PMID 26316768
- [Background] Molodecky NA, Soon IS, Rabi DM, Ghali WA, Ferris M, Chernoff G, Benchimol EI, Panaccione R, Ghosh S, Barkema HW, Kaplan GG. Increasing incidence and prevalence of the inflammatory bowel diseases with time, based on systematic review. Gastroenterology. 2012 Jan;142(1):46-54.e42; quiz e30. doi: 10.1053/j.gastro.2011.10.001. Epub 2011 Oct 14. PMID 22001864
- [Background] Bernstein CN, Eliakim A, Fedail S, Fried M, Gearry R, Goh KL, Hamid S, Khan AG, Khalif I, Ng SC, Ouyang Q, Rey JF, Sood A, Steinwurz F, Watermeyer G, LeMair A; Review Team:. World Gastroenterology Organisation Global Guidelines Inflammatory Bowel Disease: Update August 2015. J Clin Gastroenterol. 2016 Nov/Dec;50(10):803-818. doi: 10.1097/MCG.0000000000000660. No abstract available. PMID 27741097
- [Background] Tozun N, Atug O, Imeryuz N, Hamzaoglu HO, Tiftikci A, Parlak E, Dagli U, Ulker A, Hulagu S, Akpinar H, Tuncer C, Suleymanlar I, Ovunc O, Hilmioglu F, Aslan S, Turkdogan K, Bahcecioglu HI, Yurdaydin C; Members of the Turkish IBD Study Group. Clinical characteristics of inflammatory bowel disease in Turkey: a multicenter epidemiologic survey. J Clin Gastroenterol. 2009 Jan;43(1):51-7. doi: 10.1097/MCG.0b013e3181574636. PMID 18724251
- [Background] Cosnes J, Gower-Rousseau C, Seksik P, Cortot A. Epidemiology and natural history of inflammatory bowel diseases. Gastroenterology. 2011 May;140(6):1785-94. doi: 10.1053/j.gastro.2011.01.055. PMID 21530745
- [Background] Ardizzone S, Bianchi Porro G. Inflammatory bowel disease: new insights into pathogenesis and treatment. J Intern Med. 2002 Dec;252(6):475-96. doi: 10.1046/j.1365-2796.2002.01067.x. PMID 12472908
- [Background] Lang A, Salomon N, Wu JC, Kopylov U, Lahat A, Har-Noy O, Ching JY, Cheong PK, Avidan B, Gamus D, Kaimakliotis I, Eliakim R, Ng SC, Ben-Horin S. Curcumin in Combination With Mesalamine Induces Remission in Patients With Mild-to-Moderate Ulcerative Colitis in a Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2015 Aug;13(8):1444-9.e1. doi: 10.1016/j.cgh.2015.02.019. Epub 2015 Feb 24. PMID 25724700
- [Background] Hanai H, Iida T, Takeuchi K, Watanabe F, Maruyama Y, Andoh A, Tsujikawa T, Fujiyama Y, Mitsuyama K, Sata M, Yamada M, Iwaoka Y, Kanke K, Hiraishi H, Hirayama K, Arai H, Yoshii S, Uchijima M, Nagata T, Koide Y. Curcumin maintenance therapy for ulcerative colitis: randomized, multicenter, double-blind, placebo-controlled trial. Clin Gastroenterol Hepatol. 2006 Dec;4(12):1502-6. doi: 10.1016/j.cgh.2006.08.008. Epub 2006 Nov 13. PMID 17101300
- [Background] Sabzevary-Ghahfarokhi M, Soltani A, Luzza F, Larussa T, Rahimian G, Shirzad H, Bagheri N. The protective effects of resveratrol on ulcerative colitis via changing the profile of Nrf2 and IL-1beta protein. Mol Biol Rep. 2020 Sep;47(9):6941-6947. doi: 10.1007/s11033-020-05753-4. Epub 2020 Sep 4. PMID 32888128
- [Background] Nunes S, Danesi F, Del Rio D, Silva P. Resveratrol and inflammatory bowel disease: the evidence so far. Nutr Res Rev. 2018 Jun;31(1):85-97. doi: 10.1017/S095442241700021X. Epub 2017 Dec 1. PMID 29191255
- [Background] Sadeghi N, Mansoori A, Shayesteh A, Hashemi SJ. The effect of curcumin supplementation on clinical outcomes and inflammatory markers in patients with ulcerative colitis. Phytother Res. 2020 May;34(5):1123-1133. doi: 10.1002/ptr.6581. Epub 2019 Dec 4. PMID 31802559